CLINICAL TRIAL: NCT05306860
Title: Investigation of the Relationships and Clinical Parameters Between IL-6, IL-17 and IL-35 Levels in the Gingival Crevicular Fluid of Individuals With Grade B-C Stage III-IV Periodontitis
Brief Title: IL-6, IL-17 and IL-35 Levels in the Gingival Crevicular Fluid of Patients With Periodontitis and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Müge Ergün, PhD Student, Istanbul University
Other Study IDs: 679620
Record Dates: First submitted 2022-01-24; First posted 2022-04-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Periodontitis
Keywords: periodontitis; healthy gingiva; stage III; stage IV; grade b; grade c
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Biospecimen Retention: Samples Without DNA — Gingival Crevicular Fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grade B-C stage III-IV periodontitis group: Grade B-C stage III-IV periodontitis group Grade B: Moderate Moderate bone loss is observed compared to biofilm and % Root Bone Loss/age 0.25 to 1.0 is determined as grade B.
  Stage III: Severe Consisted of individuals with interdental AL ≥5 mm, radiographic bone lose extending to middle or apical third of the root, PD≥6 mm and tooth loss due to periodontitis of ≤4.
  Grade C: Rapid Rapid bone loss is observed compared to biofilm and % Root Bone Loss/age >1.0 is determined as grade C.
  Stage IV:Advanced Consisted of individuals with interdental AL ≥5 mm, radiographic bone lose extending to middle or apical third of the root, PD≥6 mm and tooth loss due to periodontitis of ≥5. Need for complex rehabilition due to: Masticatory dysfunction, Secondary occlusal trauma(tooth mobility degree ≥2) Severe ridge defect,Bite collapse, drifting, flaring. Less than 20 remaining teeth (10 opposing pairs)
  Interventions: Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis (periodontitis, healthy)
- Healthy control group: Consisted of individuals with clinically healthy gingiva on an intact periodontium who had a BOP score less than 10% and PD≤3mm, showed no attachment loss or radiographic bone loss.
  Interventions: Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis (periodontitis, healthy)

INTERVENTIONS:
Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis (periodontitis, healthy) — No intervention was applied to the groups the samples will be collected in terms of the diagnosis (periodontitis, healthy)

SUMMARY:
Periodontitis is an inflammatory disease characterized by periodontal tissue destruction caused by bacterial infection. The immune response plays an important role in the progression of periodontitis. The disease process starts with periodontopathogens in dental plaque, and tissue destruction is mainly caused by the immune response of the host to the etiological microorganism and cytokine profile through various inflammatory cytokines. The cytokine response, which plays a critical role in the pathogenesis of periodontal disease, determines the progression of the disease.

Evaluation of the effects of IL-6, IL-17 and IL-35 levels in the gingival crevicular fluid on periodontal disease together with clinical parameters has been the basis of our study. This study consists of individuals with grad B-C stage III-IV periodontitis and healthy individuals, which is the subtitle of Periodontal and Periimplant Diseases and Conditions in the classification renewed in 2017.

It is aimed to examine the changes and possible correlations in IL-6, IL-17, IL-35 levels as a result of biochemical examination of the samples taken from the gingival crevicular fluid. In our study, according to the new classification of 2017, gingival crevicular fluid samples collected from individuals with grade B-C stage III-IV periodontal disease and healthy individuals under appropriate conditions and techniques were measured for IL-6, IL-17 and IL-35 by enzymatic immunosorbent test (ELISA). It aims to investigate the negative/positive correlations and compare the increases-decreases.

DETAILED DESCRIPTION:
IL-35 is a next-generation signaling molecule belonging to the IL 12 cytokine family. It is produced by T-regulatory cells (Treg) consisting of the Α chain (p35). Recent studies have shown that IL-35 is an anti-inflammatory cytokine. It suppresses the immune response through Treg expansion and suppression of Th17 cell growth.

Interleukin-17 (IL-17) is a proinflammatory cytokine secreted by T-17 cells. It is a potent activator of neutrophils as it regulates G-CSF and receptor and chemokine expression. Its increased level has been documented in chronic periodontitis. In the presence of P. gingivalis, an increase in IL-17 and IL-23 is observed. Although periodontal infection (P. gingivalis) induces IL-17, a protective role of IL-17 against bone resorption has also been suggested. IL-17 produces IL-6, IL-8 by affecting fibroblasts.

IL-6 is produced by many cells in response to LPS and has both pro-inflammatory and anti-inflammatory roles. It is involved in inflammatory, regenerative, metabolic and neural processes. IL-6 level has been investigated in different studies in serum, saliva and gingival sulcus fluids. Studies with increased IL-6 levels in the gingival groove fluid in chronic periodontitis and studies with significant decreases in serum after nonsurgical treatment of chronic periodontitis have been reported. However, there are also studies that do not show a significant difference in the levels of various cytokines in the saliva of chronic periodontitis and healthy individuals.

Clinical measurements include Plaque Index (PI), Gingival Index (GI), Bleeding on Probing (BOP), Probing Depth (PD), Clinical attachment level (CAL), Gingival margin position (DKK), and Mobility parameters. Measurements will be recorded from six different points of all teeth by the same investigator with a Williams-type periodontal probe (Hu-Friedy, USA).

1. Healthy control groups:

   Consisted of individuals with clinically healthy gingiva on an intact periodontium who had a BOP score less than 10% and PD≤3mm, showed no attachment loss or radiographic bone loss.
2. Grade B-C / Stage III-IV periodontitis groups:

Grade B: Moderate rate of progression Moderate bone loss is observed compared to biofilm and % Root Bone Loss/age 0.25 to 1.0 is determined as grade B.

Stage III: Severe periodontitis with potential for additional tooth loss Consisted of individuals with interdental AL ≥5 mm, radiographic bone lose extending to middle or apical third of the root, PD≥6 mm and tooth loss due to periodontitis of ≤4.

Grade C: Rapid rate of progression Rapid bone loss is observed compared to biofilm and % Root Bone Loss/age >1.0 is determined as grade C.

Stage IV:Advanced periodontitis with extensive tooth loss and potential for loss of dentition Consisted of individuals with interdental AL ≥5 mm, radiographic bone lose extending to middle or apical third of the root, PD≥6 mm and tooth loss due to periodontitis of ≥5. Need for complex rehabilition due to: Masticatory dysfunction, Secondary occlusal trauma(tooth mobility degree ≥2) Severe ridge defect,Bite collapse, drifting, flaring. Less than 20 remaining teeth (10 opposing pairs)

Periodontitis Group:

* 18-65 years old
* Not having any systemic disease (diseases that do not affect the periodontal status)
* Non-smoker
* Have not received antibiotic treatment and/or used immunosuppressant medication in the last 6 months
* Have not received any periodontal treatment before
* No pregnancy and breastfeeding status
* Not using any medication regularly
* Having at least 20 teeth
* Those with grade B-C stage III-IV periodontal disease according to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions

Healthy Group:

In patients who applied to Istanbul University Faculty of Dentistry, Department of Periodontology, periodontally healthy individuals who do not meet the above disease criteria, who do not have a history of periodontitis in any way, will be included in the study.

Samples of paper strips (Periopaper®, Proflow Inc., Amitiyville, NY, USA) placed in the gingival crevicular will be placed in eppendorf tubes for laboratory examination in the session 1 week after the exact periodontal status is determined by periodontal measurements. Samples will be taken from areas with the deepest probing depth. While obtaining gingival crevicular fluid samples, the area will be isolated with cotton pads, the microbial dental plaque on the tooth will be removed with cotton pellets, and a short-term drying process will be performed with air freshener from a distance of 20 cm at a right angle. Then, standard absorbent 2x8 mm paper strips will be placed from the approximal regions to the entrance of the crevicular with slight resistance and left for 30 seconds, then each paper strip will be placed in the same eppendorf tube for each patient and stored at -80°C. (New brunswick scientific ultra low temperature freezer). Samples will be taken from 4 teeth in each patient. In case of bleeding in the gingival crevicular during sample collection, the paper strip will be discarded. The samples will be isolated from the gingival crevicular with the help of absorbent paper strips (Periopaper®, Proflow Inc., Amitiyville, NY, USA) and biochemical analyzes will be made in the samples by ELISA method in accordance with the protocols included in the kit.

Descriptive data obtained in the study will be given as Mean ± Standard Deviation (median (min-max) for each group. Testing the Normality Assumption with Hypothesis Testing, Hypothesis Testing will be analyzed with Kolmogorov - Smirnov or Shapiro-Wilk tests.

The mean differences for each group in comparisons for the two groups in the analyses; t-test in independent groups in cases where the data show normal distribution, in cases where the data do not show normal distribution; Mann-Whitney U test will be used.

In more than two groups, One Way ANOVA will be used in cases where the data are normally distributed; Multiple comparisons will be made with the Tukey test. In cases where the data do not show normal distribution, Kruskal-Wallis H test will be analyzed, and multiple comparisons will be analyzed with the Non-Parametric S-N-K Method (Student Newman-Keuls Test). Statistical significance will be considered as p< 0.05 and two-way.

According to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions, an average of 11 units difference between the results obtained from interleukin biomarkers in the group of individuals with grade B-C stage III-IV periodontitis and healthy individuals, and a minimal sample to find the estimated 15-unit standard deviation significant size (assuming Type I error 5%, Type II error 20% assuming Power 0.80): 30 people for each group. Considering the wrong samples, 30+30 people will be taken into each group (30 healthy controls, 30 Periodontitis cases).

ELIGIBILITY:
Inclusion Criteria for grade B-C stage III-IV periodontitis group:

* 18-65 years old
* Not having any systemic disease (diseases that do not affect the periodontal status)
* Non-smoker
* Have not received antibiotic treatment and/or used immunosuppressant medication in the last 6 months
* Have not received any periodontal treatment before
* No pregnancy and breastfeeding status
* Not using any medication regularly
* Having at least 20 teeth
* Those with grade B-C stage III-IV periodontal disease according to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions

Inclusion Criteria for periodontal healthy group:

•In patients who applied to Istanbul University Faculty of Dentistry, Department of Periodontology, periodontally healthy individuals who do not meet the above disease criteria, who do not have a history of periodontitis in any way, will be included in the study. Consisted of individuals with clinically healthy gingiva on an intact periodontium who had a BOP score less than 10% and PD≤3mm, showed no attachment loss or radiographic bone loss.

Exclusion Criteria:

* Those with systemic modifying disease affecting periodontal status
* Smoker
* Have received antibiotic therapy or immunosuppressive therapy in the last 6 months
* Previously received periodontal treatment in the last 6 months
* Pregnancy and breastfeeding status
* Regular use of drugs that will affect systemic health

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In our study, individuals who have Grade B-C stage III-IV periodontal disease according to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions and individuals who have healthy gingiva will be selected.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Measurement of GCF samples | GCF samples were collected after first week of clinical periodontal measurement. GCF was obtained using paper strips from the deepest gingival groove.
  Measurement of IL-6, IL-17, IL-35 levels in GCF in grade B-C stage III-IV periodontitis individuals.

SECONDARY OUTCOMES:
Measurement of GCF samples | GCF samples were collected after first week of clinical periodontal measurement. GCF was obtained using paper strips from the deepest gingival groove.
  Measurement of IL-6, IL-17, IL-35 levels in GCF with systemically-periodontally healthy (H) individuals

CONTACTS AND LOCATIONS:
Overall Officials: Emine Çifcibaşı, Assoc.Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only clinical istatical analyses and GCF samples analyses will be shared.

REFERENCES:
- [Result] Cekici A, Kantarci A, Hasturk H, Van Dyke TE. Inflammatory and immune pathways in the pathogenesis of periodontal disease. Periodontol 2000. 2014 Feb;64(1):57-80. doi: 10.1111/prd.12002. PMID 24320956
- [Result] Batool H, Nadeem A, Kashif M, Shahzad F, Tahir R, Afzal N. Salivary Levels of IL-6 and IL-17 Could Be an Indicator of Disease Severity in Patients with Calculus Associated Chronic Periodontitis. Biomed Res Int. 2018 Feb 18;2018:8531961. doi: 10.1155/2018/8531961. eCollection 2018. PMID 29670909
- [Result] Raj SC, Panda SM, Dash M, Patnaik K, Mohanty D, Katti N, Mahapatra A, Mishra D, Praharaj K. Association of Human Interleukin-35 Level in Gingival Crevicular Fluid and Serum in Periodontal Health, Disease, and after Nonsurgical Therapy: A Comparative Study. Contemp Clin Dent. 2018 Apr-Jun;9(2):293-297. doi: 10.4103/ccd.ccd_51_18. PMID 29875576
- [Result] Taniguchi T. Cytokine signaling through nonreceptor protein tyrosine kinases. Science. 1995 Apr 14;268(5208):251-5. doi: 10.1126/science.7716517.
- [Result] Taubman MA, Yoshie H, Ebersole JL, Smith DJ, Olson CL. Host response in experimental periodontal disease. J Dent Res. 1984 Mar;63(3):455-60. doi: 10.1177/00220345840630031801. PMID 6607940
- [Derived] Altaca M, Cebesoy EI, Kocak-Oztug NA, Bingul I, Cifcibasi E. Interleukin-6, -17, and -35 levels in association with clinical status in stage III and stage IV periodontitis: a cross-sectional study. BMC Oral Health. 2024 Aug 30;24(1):1015. doi: 10.1186/s12903-024-04751-3. PMID 39215253